CLINICAL TRIAL: NCT05554289
Title: Efficacy, Safety, and Acceptability of Internet-based Cognitive Behavioral Therapy Delivered Via Smartphone for Mild-to-moderate Major Depressive Disorder: a Multi-center, Double-blind, Randomized Controlled Trial
Brief Title: Efficacy, Safety, and Acceptability of Internet-based Cognitive Behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adai Technology (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICBT2021
Record Dates: First submitted 2022-09-20; First posted 2022-09-26 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Depression
Keywords: Cognitive behavioral therapy; Cognitive bias modification; Digital therapeutics
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depression Auxiliary Intervention Treatment Software (WL-iCBT) (Experimental): Participants in this arm receive the Depression Auxiliary Intervention Treatment Software (WL-iCBT) for 8 weeks. The software employs mobile-based cognitive behavioral therapy through a smartphone interface with structured interactive multimedia content. Participants use the software once daily for 10-15 minutes, completing 56 sessions over the 8-week treatment period. The intervention consists of eight progressive modules covering rational understanding of depression, methods for regulating negative emotions, and cognitive behavioral training. The software also includes attention bias modification training through "Finding Pleasure" and "Positive Action" exercises. Following the 8-week treatment period, participants enter the 26-week observational follow-up phase with no continued intervention from the study.
  Interventions: Device: Depression Auxiliary Intervention Treatment Software (WL-iCBT)
- Placebo Control Software (WL-iHE) (Placebo Comparator): Participants in this arm receive a placebo control version of the software (WL-iHE) for 8 weeks. The control software mimics the appearance and usage pattern of the active intervention but lacks the therapeutic cognitive behavioral therapy components. Participants use the software once daily for 10-15 minutes, completing 56 sessions over the 8-week treatment period. The control software has the same user interface and time requirements as the active intervention but does not deliver the structured cognitive behavioral therapy content or attention bias modification training. Following the 8-week treatment period, participants enter the 26-week observational follow-up phase with no continued intervention from the study.
  Interventions: Device: Placebo Control Software (WL-iHE)

INTERVENTIONS:
Device: Depression Auxiliary Intervention Treatment Software (WL-iCBT) — The Depression Auxiliary Intervention Treatment Software (WL-iCBT) is a mobile application for smartphones that delivers cognitive behavioral therapy (CBT) and cognitive bias modification (CBM) through structured interactive multimedia methods, including animations, videos, audio, and interactive exercises.
  Other Names: WL-iCBT Mobile Application; Wanglinuanyang; WanderLab Nuanyang
  Arms: Depression Auxiliary Intervention Treatment Software (WL-iCBT)
Device: Placebo Control Software (WL-iHE) — The placebo control software (WL-iHE) is a mobile application that mimics the appearance and usage pattern of the active intervention software but lacks the therapeutic cognitive behavioral therapy components. The software has a similar user interface and time requirements, with participants using it once daily for 10-15 minutes, completing a total of 56 sessions over the 8-week treatment period. Unlike the active intervention, the placebo software does not deliver structured cognitive behavioral therapy content or cognitive bias modification training, instead providing general health education information without specific depression treatment techniques.
  Other Names: WL-iHE Mobile Application; Health Education Placebo Software for Depression
  Arms: Placebo Control Software (WL-iHE)

SUMMARY:
This is a prospective, randomized, multicenter, double-blind, placebo-controlled phase III trial evaluating the efficacy and safety of WL-iCBT - a smartphone-based digital therapeutic combining cognitive behavioral therapy and attention bias modification. The study enrolls 315 participants aged 18-60 with mild-to-moderate MDD (MADRS score 18-30) across 11 clinical centers in China. Participants will be randomized to receive either active WL-iCBT or placebo software for 8 weeks, followed by a 26-week observational extension phase. Primary endpoint is change in MADRS score from baseline to Week 8. Secondary endpoints include treatment response rate, remission rate, anxiety symptoms (HAMA), functional impairment (SDS), and cognitive function (PDQ-D), and Clinical Global Impression rating scale (CGI). Safety monitoring includes AE/SAE recording and device deficiency assessment. Acceptability will be assessed by device performance evaluation.

DETAILED DESCRIPTION:
This investigation is a combined study that consists of an 8-week randomized controlled trial and a 26-week extended observational follow-up. It adopts a superiority design. Participants are stratified and randomly assigned in a 1:1 ratio. They are divided into two groups. One group is the active intervention group, which uses the WL-iCBT software. This software provides structured cognitive behavioral therapy (CBT) modules and attention bias modification training. The other group is the control group, which uses a placebo software. The placebo software has a matched interface but contains non-therapeutic content.

The intervention protocol requires participants to have 56 sessions over 8 weeks. Each day, they have one session, and each session lasts for 10-15 minutes. To meet the requirements, participants need to complete at least 42 sessions. The blinding of the trial is maintained through identical device interfaces for both groups.

The assessment timeline is divided into two phases. During the core treatment phase, which lasts from Week 0 to Week 8, assessments are carried out at baseline, Week 4 (±7 days), and Week 8 (±7 days). In the 26-week extended observation phase quarterly follow-ups are conducted for relapse monitoring and long-term safety assessment.

There are key assessments in this study. The primary endpoint is the change in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score from baseline to Week 8. The secondary endpoints include the MADRS response rate, which is defined as a ≥50% improvement; the MADRS remission rate, which means a score ≤10; changes in the Hamilton Anxiety Rating Scale (HAMA); functional improvement as measured by the Sheehan Disability Scale (SDS); clinician assessments using the Clinical Global Impression-Severity (CGI-S) and Clinical Global Impression-Improvement (CGI-I); and scores on the Perceived Deficiencies of Depression Questionnaire (PDQ-D) for cognitive function.

Safety monitoring is an important part of the study. All adverse events (AE) and serious adverse events (SAE) are recorded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 27.0. Device-related adverse events are also assessed. Thyroid function is monitored through measuring thyroid-stimulating hormone (TSH) levels, and suicide risk is tracked via Item 10 of the MADRS.

The study population has specific characteristics. Participants are diagnosed with major depressive disorder (MDD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria, which are confirmed by the Mini-International Neuropsychiatric Interview (MINI) 7.0.2. Those with treatment-resistant depression, those using psychotropic medications, and those with comorbid psychiatric disorders are excluded from the study.

The statistical plan of the study involves a sample size of 315 participants, with 155 in each group, taking into account a 20% dropout rate. There are three analysis sets: the Full Analysis Set (FAS), the Per Protocol Set (PPS), and the Safety Set (SS). The primary analysis uses a mixed-model for repeated measures (MMRM) to analyze the change in MADRS scores, with a superiority margin greater than 0. This integrated design enables a comprehensive evaluation of both the acute therapeutic effects and the sustained outcomes while maintaining the integrity of the trial throughout the extended observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the trial with signed informed consent
2. Age 18-60 years (inclusive), any gender
3. Clinical diagnosis of Major Depressive Disorder (MDD) according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria, confirmed by the Mini-International Neuropsychiatric Interview (M.I.N.I.7.0.2), with either single episode or recurrent episodes without psychotic features
4. Montgomery-Asberg Depression Rating Scale (MADRS) score ≥18 and <30 at screening
5. No antidepressant medication within 2 weeks prior to screening (6 weeks for fluoxetine), and assessed by the investigator as able to maintain without antidepressant medication during the trial period
6. Education level of primary school or above, able to understand the content of assessment scales, and proficient in using smartphones

Exclusion Criteria:

1. Current clinical diagnosis meeting DSM-5 criteria for psychiatric disorders other than Major Depressive Disorder (confirmed by M.I.N.I.7.0.2)
2. Treatment-resistant depression (defined as patients who failed to respond to adequate doses and duration (at least 4 weeks at maximum recommended dose) of 2 or more antidepressants with different chemical structures)
3. History of alcohol and drug dependence
4. Pregnant or lactating women, or men or women planning pregnancy during the clinical trial period
5. Current serious physical disease, thyroid disease (thyroid stimulating hormone (TSH) exceeding the upper limit of normal at screening), or patients considered by investigators to have hypothyroidism or hyperthyroidism (at the investigator's discretion, laboratory tests meeting exclusion criteria may be rechecked once within the screening period)
6. Obvious suicidal attempt or behavior, with a score ≥4 on item 10 "Suicidal Thoughts" of the MADRS scale
7. Patients who have received other antidepressant treatments within 3 months prior to enrollment, including Chinese herbal medicine, modified electroconvulsive therapy, transcranial magnetic stimulation, biofeedback therapy, light therapy, acupuncture, and other physical or systematic psychological treatments
8. Patients who explicitly express unwillingness to participate in psychological therapy or believe psychological therapy is ineffective
9. Patients who have participated in or are currently participating in drug clinical trials within 3 months prior to screening, or in other device clinical trials within 1 month prior to screening
10. Other conditions deemed unsuitable for enrollment by the investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 315 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) Score | Week 8 (end of treatment)
  Improvement in MADRS total score 8 weeks from baseline. MADRS is a clinician-rated scale that measures the severity of depressive symptoms. The scale consists of 10 items, each rated 0-6, with a total score range of 0-60. Higher scores indicate more severe depression symptoms. A decrease in score represents improvement.

SECONDARY OUTCOMES:
MADRS Treatment Response Rate | Week 4, Week 8 (end of treatment), and Week 34 (26 weeks post-treatment)
  Proportion of participants achieving at least 50% reduction in MADRS score from baseline.
MADRS Remission Rate | Week 4, Week 8 (end of treatment), and Week 34 (26 weeks post-treatment)
  Proportion of participants achieving MADRS score ≤10, indicating remission of depression symptoms.
Change in Montgomery-Asberg Depression Rating Scale (MADRS) Score | Week 4 (end of treatment) and Week 34 (26 weeks post-treatment)
  Improvement in MADRS total score from baseline. MADRS is a clinician-rated scale that measures the severity of depressive symptoms. The scale consists of 10 items, each rated 0-6, with a total score range of 0-60. Higher scores indicate more severe depression symptoms. A decrease in score represents improvement.
Change in Hamilton Anxiety Scale (HAMA) Score | Week 4, Week 8 (end of treatment), and Week 34 (26 weeks post-treatment)
  Improvement in HAMA total score from baseline. HAMA is a 14-item scale measuring the severity of anxiety symptoms with a total score range of 0-56. Higher scores indicate more severe anxiety symptoms.
Change in Clinical Global Impression (CGI) Score | Week 4, Week 8 (end of treatment), and Week 34 (26 weeks post-treatment)
  Changes in CGI-Severity (CGI-S) score from baseline and CGI-Improvement (CGI-I) score. CGI-S rates illness severity on a 7-point scale, and CGI-I rates improvement relative to baseline on a 7-point scale. For CGI-S, lower scores indicate improvement; for CGI-I, lower scores indicate greater improvement.
Change in Sheehan Disability Scale (SDS) Score | Week 4, Week 8 (end of treatment), and Week 34 (26 weeks post-treatment)
  Improvement in SDS score from baseline. SDS assesses functional impairment in work/school, social life, and family life domains.
Change in Perceived Deficiencies of Depression Questionnaire (PDQ-D) Score | Week 4, Week 8 (end of treatment), and Week 34 (26 weeks post-treatment)
  Improvement in PDQ-D score from baseline. PDQ-D is a self-assessment questionnaire measuring cognitive deficits associated with depression, with higher scores indicating greater perceived cognitive impairment.
Incidence of Adverse Events | From randomization through Week 34 (26 weeks post-treatment)
  Number and percentage of participants experiencing adverse events, including device-related adverse events.
Device Performance Evaluation | Week 8 (end of treatment)
  Researcher assessment of the software's performance for both researcher and participant interfaces, rated on a scale of excellent, good, moderate, or poor. Device performance excellence rate is calculated as the percentage of "excellent" and "good" ratings.
Incidence of Device Defect | Week 8 (end of treatment)
  Number and percentage of participants experiencing device malfunctions and defects.

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Shenzhen Kangning Hospital, Shenzhen, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Zhumadian Second People's Hospital, Zhumadian, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shannxi
  - Chengdu Fourth People's Hospital (Chengdu Mental Health Center), Chengdu, Sichuan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunan
  - Zhejiang Provincial Tongde Hospital, Hangzhou, Zhejiang
  - Ningbo Kangning Hospital, Ningbo, Zhejiang
  - Quzhou Third Hospital, Quzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD.